CLINICAL TRIAL: NCT01019876
Title: Risk-Adapted Allogeneic Stem Cell Transplantation For Mixed Donor Chimerism In Patients With Selected Non-Malignant Diseases
Brief Title: Risk-Adapted Allogeneic Stem Cell Transplantation For Mixed Donor Chimerism In Patients With Non-Malignant Diseases
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Columbia University (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: AAAB0170; CHNY-01-509 (Other: CU)
Record Dates: First submitted 2009-11-23; First posted 2009-11-25 (Estimated); Last update posted 2024-10-31 (Actual); Status verified 2024-10

CONDITIONS: Bone Marrow Failure; Osteopetrosis; Fanconi Anemia; Severe Combined Immunodeficiency
Keywords: Bone marrow Failure; Fanconi Anemia; Severe Combined Immunodeficiency; Osteopetrosis; Allogeneic Stem Cell Transplantation; Chemotherapy; Radiation Therapy
MeSH Terms: conditions — Bone Marrow Failure Disorders; Osteopetrosis; Fanconi Anemia; Severe Combined Immunodeficiency | interventions — fludarabine; fludarabine phosphate; Cyclophosphamide; Busulfan; Alemtuzumab; Antilymphocyte Serum; thymoglobulin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Regimen A - Standard Conditioning Regimen (Active Comparator): Standard conditioning regimen for all diseases except those diseases or conditions noted in Regimen B, C and D:
  * Fludarabine (180 mg/m2 total dose)
  * Busulfan (16 mg/kg less than or equal to 4 yrs and 12.8 mg/ kg >4 yrs total dose)
  * Alemtuzumab (2mg/m2 x 1day, 6mg/m2 x 2 days, 20mg/m2 x 2days)
  Interventions: Drug: Fludarabine; Drug: Busulfan; Drug: Alemtuzumab
- Regimen B (Experimental): Includes patients with a diagnosis of: Osteopetrosis and Severe Aplastic Anemia with a history of >10 blood transfusions, or Blackfan-Diamond's anemia, or Chronic Granulomatous Disease, or Wiskott Aldrich Syndrome:
  * Cyclophosphamide (200 mg/kg total dose)
  * Fludabarine (180 mg/m2 total dose)
  * Rabbit Anti-thymocyte Globulin (8mg/kg total dose)
  Interventions: Drug: Fludarabine; Drug: Cyclophosphamide; Drug: Rabbit Anti-thymocyte Globulin
- Regimen C (Experimental): Includes patients with any one of the following speciﬁc diagnosis: Fanconi Anemia, Dyskeratosis Congenita or Schwachman Diamond Syndrome
  * Cyclophosphamide (40 mg/kg total dose)
  * Fludarabine (140 mg/m2 total dose)
  * Anti-Thymocyte Globulin (horse) (150mg/kg total dose)/TBI 450 cGy
  Interventions: Drug: Fludarabine; Drug: Cyclophosphamide; Drug: Horse Anti-thymocyte Globulin
- Regimen D (Experimental): Includes patients with the following speciﬁc diagnosis of: Severe Combined Immune Deﬁciency Syndrome with no evidence of host NK function (will receive Regimen A) and matched related donor
  * Cyclophosphamide (30 mg/kg total dose)
  * Fludarabine (90 mg/m2 total dose)
  * Rabbit anti-thymocyte globulin (Thymoglobulin)(TMG)**(8 mg/kg total dose)
  TMG only in family haploidentical and unrelated donors
  Interventions: Drug: Fludarabine; Drug: Cyclophosphamide; Drug: Rabbit Anti-thymocyte Globulin

INTERVENTIONS:
Drug: Fludarabine
  Other Names: Fludara®
Drug: Cyclophosphamide
  Other Names: Cytoxan®
  Arms: Regimen B; Regimen C; Regimen D
Drug: Busulfan
  Other Names: Busulfex®
  Arms: Regimen A - Standard Conditioning Regimen
Drug: Alemtuzumab
  Other Names: Campath®
  Arms: Regimen A - Standard Conditioning Regimen
Drug: Rabbit Anti-thymocyte Globulin
  Other Names: TMG; Thymoglobulin
  Arms: Regimen B; Regimen D
Drug: Horse Anti-thymocyte Globulin
  Other Names: ATG; Lymphocyte Immune Globulin
  Arms: Regimen C

SUMMARY:
This study proposes the use of a reduced intensity chemotherapy/radiation therapy regimen followed by stem cell transplantation, as compared to standard ablative chemotherapy regimens associated with stem cell transplantation, in a population of patients with non-malignant diseases (non-cancer). Eligible patients will have a non-malignant disease in one of the following four strata: bone marrow failure syndromes, immunodeﬁciencies, inborn errors of metabolism, or histiocytoses. Patients will be assigned to therapy according to diagnosis. Patients will be stratiﬁed by disease into one of four strata and treatment regimens will be based on speciﬁc disease criteria and conditions. Although these diseases are non-malignant in name, they are often malignant by nature of the disease progression, treatment and associated complications.

DETAILED DESCRIPTION:
This treatment program proposes the use of a reduced intensity chemotherapy regimen, which has been shown to be effective for inducing remission and cure in these diseases. Studies have shown that the use of non-myeloablative chemotherapy regimens have resulted in 75-100% engraftment (replacement of the recipient bone marrow with the donor bone marrow), and signiﬁcantly reduced transplant related complications as compared to the standard myeloablative chemotherapy regimens.

ELIGIBILITY:
Inclusion Criteria

Patients must meet the eligibility criteria for organ function regardless of diagnosis:

* Age < 30 or = 30 years of age
* Adequate renal function defined as serum creatinine < or = 1.5 x normal, or creatinine clearance or radioisotope glomerular filtration rate (GFR) > or =40 ml/min/m2 or >60 ml/min/1.73 m2 or an equivalent GFR as determined by the institutional normal range
* Adequate liver function defined as serum glutamic oxaloacetic transaminase (SGOT)(Aspartate transaminase (AST)) or serum glutamic-pyruvic transaminase (SGPT) (alanine aminotransferase (ALT)) < 5.0 x normal
* Adequate cardiac function defined as shortening fraction of > or = 28% by echocardiogram, or ejection fraction of > or = 48% by radionuclide angiogram or echocardiogram
* Adequate pulmonary function defined as asymptomatic or, if symptomatic, carbon monoxide diffusing capacity test (DLCO) >45% of predicted (corrected for hemoglobin level). If unable to obtain pulmonary function test, O2 saturation >85% in room air.

Bone Marrow Failure Syndromes

Patients with the following diagnoses are eligible:

Severe Aplastic Anemia:

* Hypocellular bone marrow biopsy (<25% cellularity) and 2/3 of the following (at diagnosis or nadir):
* Absolute Neutrophil Count (ANC) <200/mm3,
* Platelets <20,000/mm3
* Reticulocyte count <60,000/mm3

Fanconi Anemia:

* Abnormal clastogenic studies (all patients) Severe Congenital Neutropenia (Kostmann's Syndrome) Amegakaryocytic Thrombocytopenia
* Severe thrombocytopenia (< or =20,000/mm3) at diagnosis
* Severe depletion of megakaryocytes on bone marrow aspirate (< or =25% normal)

Diamond-Blackfan Anemia:

* Corticosteroid dependent for > 6 months OR Transfusion dependent OR refractory acquired pure red cell aplasia.

Infantile Osteopetrosis Schwachman-Diamond Syndrome Dyskeratosis Congenita Other bone marrow failure syndromes at discretion of co-principal investigators All BM failure patients must have BM bx within 2 weeks prior to starting therapy to confirm disease status

Immunodeficiencies:

* SCIDS, all subtypes
* Combined Immunodeficiency Syndrome
* Wiskott-Aldrich Syndrome
* Chronic Granulomatous Disease
* Chediak-Higashi Syndrome
* Leukocyte Adhesion Deficiency
* Other immunodeficiencies at discretion of co-principal investigators

Inborn Errors of Metabolism (IEOM):

Transplant is recommended for the following disorders:

* Hurler syndrome (alpha-L-iduronidase deficiency, MPS-I), preferably before age 24 months
* Maroteaux-Lamy syndrome (galactosamine-4-sulfatase deficiency,MPSVI)
* Sly syndrome (beta-glucuronidase deficiency, MPS-VII)
* Globoid cell leukodystrophy (galactocerebrosidase deficiency), with careful attention to neurologic status in the infantile form
* Metachromatic leukodystrophy (arylsulfatase A deficiency),juvenile or adult onset form; late infantile MLD only if pre-symptomatic
* Childhood-onset X-linked adrenoleukodystrophy (X-ALD), at initial signs of neuropsychological deterioration, with dietary modification prior to transplant
* Fucosidosis (fucosidase deficiency)
* Mannosidosis
* Aspartylglucosaminuria
* Niemann-Pick Disease Type B (acid sphingomyelinase deficiency)
* Other diagnoses may be considered at the discretion of the co-principal investigators

Transplant is not recommended for Hunter syndrome (iduronate sulfatase deficiency), Sanfilippo syndrome Type A (heparan N-sulfatase deficiency), Sanfilippo syndrome Type B (-N-acetyl-transferase deficiency), Sanfilippo syndrome Type C (-acetyltransferase deficiency), Sanfilippo syndrome Type D (-acetylglucosamine-6-sulfatase deficiency), Morquio syndrome (galactose-6-sulfatase deficiency); or Niemann-Pick disease Type A or C.

For X-ALD patients greater than 5 years of age, IQ >80 is required. For other patients greater than 5 years of age, IQ > 70 is required.

For patients less than 5 years of age, the developmental quotient or clinical neurodevelopmental examination should demonstrate potential for stabilization at a level of functioning where continuous life support (e.g. mechanical ventilation) would not be predicted to be required in the year following transplantation.

For Gaucher disease (glucocerebrosidase deficiency) Type I (non-neuropathic), the primary therapy is enzyme replacement, but allogeneic stem cell transplant has been used effectively.

Histiocytoses:

* Hemophagocytic Lymphohistiocytosis (HLH)
* Familial Erythrophagocytic Lymphohistiocytosis
* Langerhans Cell Histiocytosis
* Patients with multi-system disease whose initial disease is stable or progressive after minimum 6 weeks of appropriate therapy, OR patients with recurrent multi-system disease.
* Malignant Histiocytosis
* All histiocytic patients must have BM bx within 2 weeks prior to starting therapy to confirm disease status

Other non-malignant diseases not listed above may be eligible if deemed appropriate by the co-principal investigators.

Max Age: 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 38 (Actual)
Dates: Start 2002-09 (Actual); Primary Completion 2021-09-07 (Actual); Study Completion 2021-09-07 (Actual)

PRIMARY OUTCOMES:
Number of participants with Adverse Events | Up to 2 years
  The number of participants with adverse events as assessed by National Cancer Institute (NCI) Common Terminology Criteria Adverse Events (CTCAE - Version 4.0)

SECONDARY OUTCOMES:
Risk of disease progression | Up to 1 year
  To determine the risk of disease progression (including neuropsychological deterioration in patients with metabolic non-malignant diseases) following a Flu/CY or Bu/Flu based conditioning regimen.
Immune reconstitution | Up to 1 year
  Titers of immune cells (T cells, B cells, and NK cells) from peripheral blood will be measured following a Flu/CY or Bu/Flu based conditioning regimen and AlloSCT in patients with selected non-malignant diseases.
Incidence of graft versus host disease (GVHD) | Up to 1 year
  Incidence of GVHD in participants following a Flu/Cy or Bu/Flu based conditioning regimen.
Metabolic/Immune reconstitution | Up to 1 year
  To determine metabolic/immune (gene/protein) reconstitution by standard biochemical/PCR assays in patients.

CONTACTS AND LOCATIONS:
Overall Officials: James Garvin, MD, PhD, Principal Investigator — Columbia University
Locations (1):
- Columbia University Medical Center, New York, New York, United States